CLINICAL TRIAL: NCT06626178
Title: ARtificial Intelligence for heAlth and Prevention of Smoking-related Diseases
Brief Title: Development of an Artificial Intelligence Model for the Identification and Prevention of Smoking-related Diseases.
Acronym: ARIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Muriana Piergiorgio, Medical Doctor, Scientific Institute San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CET 288-2024
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer Screening Program; Artificial Intelligence (AI)
Keywords: CT scan low-dose; Artificial Intelligence; High-risk sucjects; Lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, X-Ray Computed; Radionuclide Imaging; Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: In the study are considered 4 different cohorts. Lung cancer patients diagnosed outside screening and treated at San Raffaele Hospital; smokers and former smokers aged over 50 years old at high risk for lung cancer, cardiovascular diseases and chronic obstructive pulmonary disease (COPD); subjects enrolled in previous screening cohorts in this Institute, which presented a computed tomography (CT) with the presence of lung nodules >4 mm and to conclude, subjects enrolled in previous screening cohorts in this Institute, which presented a negative computed tomography (CT).
Masking Description: No blinding in this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-risk screening subjects (Experimental): Ever and former male and female smokers aged over 50 years old at high risk for lung cancer, cardiovascular diseases and chronic obstructive pulmonary disease (COPD).
  Additional procedures for this group:
  * Spirometry
  * Nurse evaluation
  * Epidemiological questionnaire, Quality of Life (QoL) questionnaires
  * Smoking cessation program
  * Cardiovascular primary prevention
  * measurement of carbon monoxide (CO)
  * Blood storage
  * Computed tomography (CT) scan low-dose
  Interventions: Diagnostic Test: Computed tomography (CT) scan low dose; Procedure: Blood sampling; Other: Spirometry; Other: Questionnaires; Other: Smoking cessation program; Other: Carbon monoxide measurment; Other: Cardiovascular primary prevention
- Previous positive high-risk screening subjects (Experimental): Subjects enrolled in previous screening cohorts in this Institute with the presence of lung nodules >4 mm. Additional procedure for this group: Computed tomography (CT) scan low-dose
  Interventions: Diagnostic Test: Computed tomography (CT) scan low dose; Other: Smoking cessation program
- Previous negative high-risk screening subjects (No Intervention): Subjects enrolled in previous screening cohorts in this Institute with negative computed tomography (CT) scan. No additional procedures for this group.
- Lung cancer patients (Experimental): Lung cancer patients diagnosed outside screening and treated at San Raffaele Hospital. Additional procedures for this group: biobank tissue and blood storage.
  Interventions: Procedure: Blood sampling; Procedure: Tissue sampling (lung)

INTERVENTIONS:
Diagnostic Test: Computed tomography (CT) scan low dose — The radiological investigation will be done with multi-detector-row (64 or more) computed tomography (CT) scanners at low-dose protocol. The low-dose spiral CT consists of a CT study of the chest, without the need for injection of contrast medium, characterized by less radio exposure than the standard CT of the chest with high sensitivity in detecting pulmonary nodules.
  Arms: High-risk screening subjects; Previous positive high-risk screening subjects
Procedure: Blood sampling — Peripheral venous blood sampling (20 ml)
  Arms: High-risk screening subjects; Lung cancer patients
Procedure: Tissue sampling (lung) — sampling of tumor and healthy tissue during surgery
  Arms: Lung cancer patients
Other: Spirometry — Spirometry measurement using spirometer
  Arms: High-risk screening subjects
Other: Questionnaires — Compilation of epidemiological questionnaire, quality of life questionnaires
  Arms: High-risk screening subjects
Other: Smoking cessation program — Study guarantee valid support for quitting smoking, which for a smoker is a more effective intervention to reduce the risk of developing lung cancer, myocardial infarction and other smoking-related diseases
  Arms: High-risk screening subjects; Previous positive high-risk screening subjects
Other: Carbon monoxide measurment — Measurment of Carbon monoxide (CO)
  Arms: High-risk screening subjects
Other: Cardiovascular primary prevention — Intervention done in order to find the presence of coronary calcifications
  Arms: High-risk screening subjects

SUMMARY:
The study is an interventional pilot study. The study is designed to be monocentric and it presents additional procedues.

DETAILED DESCRIPTION:
Interventional pilot study, single-center with additional procedures, such as completion of EORTC-QLQ-LC29, EORTC-QLQ-C30 questionnaires, motivational test, Fagestrom test, anamnestic questionnaire, spirometry, measurement of carbon monoxide, Low-dose spiral computed tomography without contrast medium, peripheral venous blood sampling for a volume of 20 ml.

The study has the main objective of traininig and validate a reliable and unbiased Artificial Intelligence (AI) algorithm that detects the presence of nodules and differentiates between malignant or benign tumor types.

The study considers patients with suspected diagnosis or with a dignosis of lung cancer, smokers and former smokers over 50 years of age at high risk of lung cancer and subjects enrolled in previous screening cohorts at this Institute.

ELIGIBILITY:
High-risk screening subjects

Inclusion Criteria:

* Age >= 50 years old
* Active smokers
* Former smokers (from no more than 15 years)
* Pack/year >20
* Risk-prediction model from Prostate, Lung, Colorectal, and Ovarian study (PLCOm2012) >1.2%
* Provision and signature of informed consent

Exclusion Criteria:

* Previous or concurrent neoplastic disease, excluding skin cancers
* Cognitive or other problems that could hinder the collection of informed consent
* Severe pulmonary or extra pulmonary disease
* Previous low-dose computed tomography (CT) scan in the past 12 months

Previous high-risk positive screening subjects

Inclusion Criteria:

* Subjects enrolled in previous lung cancer screening with the presence of lung nodules >4 mm and candidate to additional computed tomography (CT)
* Signed informed consent

Exclusion Criteria:

- None

Previous high-risk negative screening subjects

Inclusion Criteria:

* Subjects enrolled in previous lung cancer screening in this Institute with negative computed tomography (CT)
* Signed informed consent

Exclusion Criteria:

- None

Lung Cancer patients

Inclusion Criteria:

* Patients with diagnosis or suspicious diagnosis of lung cancer candidate to surgical treatment or already submitted to it
* Patients with diagnosis of lung cancer treated with surgical resection
* Signed informed consent

Exclusion Criteria:

* computed tomography (CT) scans not available at San Raffaele Hospital
* Previous neoadjuvant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2840 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Creation of Artificial Intelligence (AI) algorithm | from enrollment to 48 months
  To train and validate a reliable and unbiased Artificial Intelligence (AI) algorithm that detects the presence of nodules and differentiates between malignant or benign tumor types.
  AUC (Area Under the Curve) values, expressed as mean and standard deviation (SD), comparing the ability in detecting the presence of nodules and differentiating the malignancy or benignity of a radiologist versus an AI algorithm, both trained on the same patient group.

SECONDARY OUTCOMES:
Multimodal program | from enrollment to 48 months
  Develop a multimodal program to enhance the prevention and the early detection of multiple smoking-related diseases Presence and absence of lung nodules > 4 mm with computed tomography (CT) scan

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute Ospedale San Raffaele, Milan, Italy